CLINICAL TRIAL: NCT02741869
Title: Photodisinfection for the Decolonization of Staphylococcus Aureus in Hemodialysis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator moved locations.
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HD.SA-1
Record Dates: First submitted 2016-02-29; First posted 2016-04-18 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Staphylococcus Aureus Infection; MSSA Colonization
Keywords: Staphylococcus aureus; nare carriage
MeSH Terms: conditions — Staphylococcal Infections | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental): This is a single arm, open label study. Subjects who meet eligibility criteria will be treated with photodisinfection therapy (MRSAid™).
  Interventions: Device: photodynamic therapy (Ondine: MRSAid™)

INTERVENTIONS:
Device: photodynamic therapy (Ondine: MRSAid™) — Photodisinfection using MRSAid™ for the decolonization of S. aureus in hemodialysis patients
  Other Names: MRSAid™

SUMMARY:
The purpose of the study is to evaluate whether PDT (MRSAid™) is effective in eradicating SA from hemodialysis patients who are known to harbor this organism inside their nose.

DETAILED DESCRIPTION:
This is a medical research study is to eliminate Staphylococcus aureus (SA) (decolonization) from nares of patients who are colonized with this organism. Bacterial colonization of the anterior nares (inside of the nose) is believed to play an important role in the development of infection of central venous catheter, such as the line used for hemodialysis, and subsequent bloodstream infection.

Photodynamic therapy (PDT) has been shown to be lethal against all classes of microorganisms: Gram-positive and, Gram-negative bacteria, fungi (fungus), viruses, parasites and even spores. In addition to the antimicrobial effects PDT also demonstrates an anti-inflammatory effect.

The objective of this study is to evaluate the efficacy of PDT in nasal decolonization of S. aureus in hemodialysis patients

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to provide written informed consent. (If the patient is unable to provide written informed consent, the patient's legally accepted representative may provide written consent as approved by institution-specific guidelines)
* Age ≥ 18
* Currently undergoing hemodialysis and has hemodialysis catheter in-situ
* Positive SA culture from anterior nare within 2 weeks of enrollment.
* Have had no antibacterial therapy for any reason within the previous 7 days
* Patient is willing and able to return for treatment and evaluation procedures scheduled throughout the course of this clinical study

Exclusion Criteria:

* Patient has taken antibiotics in the last 7 days
* Patient has taken an investigational medication in the last 30 days or is involved in a clinical study
* Women who are pregnant, nursing or of child-bearing potential and not using a medically accepted, effective method of birth control (e.g., condom, hormonal contraceptive, indwelling intrauterine device, sexual abstinence)
* Patient uses nasal medication that cannot be discontinued on the day of scheduled photodisinfection therapy.
* Patient is on oxygen via nasal cannula
* Patient has an active malignancy of any type by patient report, except for basal cell carcinoma
* Patient's surgery involves the nasal or oral cavity (e.g. repair of deviated septum)
* Patient has had surgery of the nasal tract or sinuses within the prior 3 months
* Patient has a history of moderate to severe hypersensitivity reactions to methylene blue (mild rash is not a contraindication to enrollment)
* Patient has active ulcerations of the nasal septum
* Patient has nasal polyps
* Patient has suspected or confirmed rhinosinusitis as evidenced by all three of the following:
* Sneezing
* Nasal congestion or rhinorrhea
* Patient has suspected or confirmed sinusitis
* Patient has suspected or confirmed upper respiratory infection as evidenced by at least one of the following symptoms:
* Fever of up to 38 oC.
* Sore throat, laryngitis
* Post-nasal mucus, cough
* Patient has any rapidly progressing disease or immediately life-threatening illness including acute hepatic failure, respiratory failure and septic shock
* Patient has an immunocompromising illness including known infection with human immunodeficiency virus (HIV), AIDS, hematological malignancy and bone marrow transplantation, or immunosuppressive therapy including cancer chemotherapy, medications for prevention of organ transplantation rejection, imuran and the administration of corticosteroids equivalent to or greater than 40 mg of prednisone per day administered for more than 14 days
* Patient is anticipated to receive any amount of potentially therapeutic antimicrobial therapy after collection of the pretreatment baseline culture and before administration of the study treatment
* Patient has a current urinary catheter that will not be removed or anticipation of urinary catheter placement that will not be removed during the course of study treatment. (Clarification: Intermittent straight catheterization after the study treatment is acceptable.)
* Patient has a concomitant infection requiring systemic antibiotic or antifungals at the time of assignment of patient number
* Patient has any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05 (Estimated); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
The efficacy of PDT in nasal decolonization of S. aureus in hemodialysis patients by measuring number of participants with successful decolonization of S. aureus | 1 year
  30 patients will be recruited. Success of decolonization will be determined by serial culture of nare swabs for S. aureus.

IPD SHARING:
Plan to Share IPD: No